CLINICAL TRIAL: NCT06138509
Title: Role of Peripheral Serotonin in Oculocutaneous Albinism
Brief Title: Peripheral Serotonin and Albinism
Acronym: SEPIAs
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230808; 2023-A01431-44 (Other: IDRCB Number)
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Oculocutaneous Albinism
Keywords: Oculocutaneous albinism; Peripheral serotonin; Anemia; Microcytosis; Iron deficiency
MeSH Terms: conditions — Albinism, Oculocutaneous; Anemia; Iron Deficiencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Patients with albinism aged 2 to 17 years old and followed in the MAGEC-Necker reference center (reference center for rare diseases of the skin and mucous membranes of genetic origin), during the inclusion period.
  During an initial or a follow-up consultation for patients with albinism, an additional volume of blood will be drawn during a blood sample drawn as part of routine care.
  Interventions: Other: Dosage of serotonin and metabolites; Other: Blood parameters
- Control patients: Control patients are patients who were seen at Necker-Enfants Malades Hospital during the inclusion period, in the emergency and surgical departments, and whose care required a blood test analyzed in the Necker-Enfants Malades Hospital hematology laboratory.
  These patients will be selected on their age (2 to 17 years old), and must have a normal complete blood count and CRP. Leftover blood not used by the hospital hematology laboratory will be used for study analyses.
  Interventions: Other: Dosage of serotonin and metabolites; Other: Blood parameters

INTERVENTIONS:
Other: Dosage of serotonin and metabolites — The dosages of serotonin and its metabolites will be performed by the INSERM U1016 unit at Cochin Institute.
Other: Blood parameters — The characterization of blood parameters : complete blood count (CBC), reticulocytes, C-reactive protein (CRP), iron studies (ferritin, serum iron, transferrin and transferrin saturation), hemoglobin electrophoresis, erythropoietin, will be added using standard methods at the Necker hematology laboratory if not carried out as part of the routine care.

SUMMARY:
Serotonin (5-HT or 5-hydroxytryptamine) is a monoamine primarily known for its role as a neurotransmitter in the central nervous system (CNS). However, the functions of serotonin go beyond its role in the central nervous system: different peripheral tissues have the capacity to produce and/or use serotonin locally, forming systems called "micro-serotonergic" systems. Among the peripheral roles of serotonin, previous work by the Iron and Immunity team, INSERM U1016, Institut Cochin (Paris), was able to show that serotonin has a positive role on erythropoiesis and the survival of red blood cells, and the team's ongoing work suggests that serotonin also impacts iron metabolism.

In humans and in mouse models, several studies have suggested a role for serotonin in pigmentation. In certain syndromic forms of albinism such as Hermansky Pudlak syndrome, platelet serotonin levels are reduced in connection with a decrease in dense platelet granules (delta granules): this characteristic is even part of the diagnostic criteria.

Preliminary data from the Iron and Immunity team found:

* Changes in serotonin levels in children with albinism compared to control patients,
* Changes in hemoglobin level and mean corpuscular volume (MCV) in children with albinism (towards anemia and microcytosis),
* Changes in the iron balance in children with albinism (towards iron deficiency).

The hypothesis of this research is that peripheral serotonin plays a role in the clinical and biological manifestations of oculocutaneous albinism.

DETAILED DESCRIPTION:
Serotonin (5-HT or 5-hydroxytryptamine) is a monoamine primarily known for its role as a neurotransmitter in the central nervous system (CNS). However, the functions of serotonin go beyond its role in the central nervous system: different peripheral tissues have the capacity to produce and/or use serotonin locally, forming systems called "micro-serotonergic" systems. Among the peripheral roles of serotonin, previous work by the Iron and Immunity team, INSERM U1016, Institut Cochin (Paris), was able to show that serotonin has a positive role on erythropoiesis and the survival of red blood cells, and the team's ongoing work suggests that serotonin also impacts iron metabolism.

Albinism exhibits significant clinical and genetic heterogeneity with poor genotype-phenotype correlation, and nearly 15% of patients remain without a molecular diagnosis. There is no curative treatment for albinism. Patients with albinism suffer from physical disability throughout their lives, but can also suffer from psychological disability and discrimination. These patients are also more vulnerable to the effects of climate change. The unmet clinical needs are therefore enormous.

In humans and in mouse models, several studies have suggested an unexpected role for serotonin in skin pigmentation at several levels. Transcriptomic studies revealed that the Tph1 gene, responsible for serotonin synthesis outside the CNS, as well as serotonin receptors, were expressed in melanocytic and keratinocytic cell lines. Other studies have indicated that serotonin enhances melanogenesis in three melanocyte cell lines (B16F10, SK-MEL-2, Melan-a). Finally, studies suggest that serotonin is involved in pathologies such as certain congenital dyschromias, Rett syndrome and vitiligo. In certain syndromic forms of albinism such as Hermansky Pudlak syndrome, platelet serotonin levels are reduced in connection with a decrease in dense platelet granules (delta granules): this characteristic is even part of the diagnostic criteria.

Preliminary data from the Iron and Immunity team found:

* Changes in serotonin levels in children with albinism compared to control patients,
* Changes in hemoglobin level and mean corpuscular volume (MCV) in children with albinism (towards anemia and microcytosis),
* Changes in the iron balance in children with albinism (towards iron deficiency).

The hypothesis of this research is that peripheral serotonin plays a role in the clinical and biological manifestations of oculocutaneous albinism.

The study will assess serotonin and its metabolites in the serum of patients with albinism, and compare the results with controls patients. The level of serotonin and its metabolites will be correlated with the different genotypes, and with the severity of albinism within the same genotypes.

This study also wish to explore the impact of serotonin levels in the development of anemia, microcytosis and/or iron deficiency in patients with albinism. Complete blood counts and iron studies in patients with albinism will be compare to those of control patients too.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Patients with albinism aged 2 to 17 years
* Followed in the MAGEC-Necker reference center (reference center for rare diseases of the skin and mucous membranes of genetic origin), during the inclusion period
* Information of parental authority holders of patients and patients of understanding age, and collection of consent from parental authority holders and patients.

Controls:

* Patients aged 2 to 17 years old
* Having consulted in Necker hospital during the inclusion period in the emergency and surgical services and whose care required a blood test analyzed in the hematology laboratory of the Necker hospital.
* Normal complete blood count (CBC)
* Normal C-reactive protein test (CRP)
* Absence of opposition from parental authority holders within one month of after sending the study information note.

Exclusion Criteria:

Patients:

- Inability to have a blood test

Controls:

* Abnormal blood count
* Elevation of CRP above laboratory standard

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will be recruited during a dermatology consultation at the Necker-Enfants Malades hospital. Recruitment, diagnosis of albinism and clinical, dermatological and ophthalmological characterization, as well as biological tests, will be carried out by the MAGEC reference center in Necker hospital (reference center for rare diseases of the skin and mucous membranes of genetic origin).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Level of serotonin and its metabolites in serum | Day 0
  Levels of serotonin and its metabolites in serum in children with albinism, compared with control children.

SECONDARY OUTCOMES:
Correlation between serotonin levels and molecular subtype of albinism | Day 0
  Sequencing allowing molecular characterization of albinism is an integral part of diagnosis.
Correlation between serotonin levels and severity of albinism | Day 0
  The severity of albinism : cutaneous severity is based on clinical estimation, and ophthalmological severity on visual acuity values and degree of foveal hypoplasia.
Correlation between serotonin levels and iron studies | Day 0
  Determination of ferritin, serum iron, transferrin and transferrin saturation.
Correlation between serotonin levels and hemoglobin | Day 0
  Results of complete blood count, reticulocytes, hemoglobin electrophoresis in case of microcytosis, and erythropoietin dosage.

CONTACTS AND LOCATIONS:
Overall Officials: Smail HADJ-RABIA, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Guillemette FOUQUET, MD, Study Director — Centre Hospitalier Sud Francilien (CHSF) and Cochin Institute, INSERM U1016, Team Iron and Immunity
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amireault P, Sibon D, Cote F. Life without peripheral serotonin: insights from tryptophan hydroxylase 1 knockout mice reveal the existence of paracrine/autocrine serotonergic networks. ACS Chem Neurosci. 2013 Jan 16;4(1):64-71. doi: 10.1021/cn300154j. Epub 2012 Nov 7. PMID 23336045
- [Background] Yabut JM, Crane JD, Green AE, Keating DJ, Khan WI, Steinberg GR. Emerging Roles for Serotonin in Regulating Metabolism: New Implications for an Ancient Molecule. Endocr Rev. 2019 Aug 1;40(4):1092-1107. doi: 10.1210/er.2018-00283. PMID 30901029
- [Background] Fouquet G, Coman T, Hermine O, Cote F. Serotonin, hematopoiesis and stem cells. Pharmacol Res. 2019 Feb;140:67-74. doi: 10.1016/j.phrs.2018.08.005. Epub 2018 Aug 11. PMID 30107202
- [Background] English KB, Wang ZZ, Stayner N, Stensaas LJ, Martin H, Tuckett RP. Serotonin-like immunoreactivity in Merkel cells and their afferent neurons in touch domes from the hairy skin of rats. Anat Rec. 1992 Jan;232(1):112-20. doi: 10.1002/ar.1092320112. PMID 1536455
- [Background] Johansson O, Liu PY, Bondesson L, Nordlind K, Olsson MJ, Lontz W, Verhofstad A, Liang Y, Gangi S. A serotonin-like immunoreactivity is present in human cutaneous melanocytes. J Invest Dermatol. 1998 Dec;111(6):1010-4. doi: 10.1046/j.1523-1747.1998.00460.x. PMID 9856809
- [Background] Lee HJ, Park MK, Kim SY, Park Choo HY, Lee AY, Lee CH. Serotonin induces melanogenesis via serotonin receptor 2A. Br J Dermatol. 2011 Dec;165(6):1344-8. doi: 10.1111/j.1365-2133.2011.10490.x. Epub 2011 Oct 17. PMID 21711335
- [Background] Slominski A, Pisarchik A, Semak I, Sweatman T, Wortsman J, Szczesniewski A, Slugocki G, McNulty J, Kauser S, Tobin DJ, Jing C, Johansson O. Serotoninergic and melatoninergic systems are fully expressed in human skin. FASEB J. 2002 Jun;16(8):896-8. doi: 10.1096/fj.01-0952fje. Epub 2002 Apr 23. PMID 12039872
- [Background] Slominski A, Pisarchik A, Zbytek B, Tobin DJ, Kauser S, Wortsman J. Functional activity of serotoninergic and melatoninergic systems expressed in the skin. J Cell Physiol. 2003 Jul;196(1):144-53. doi: 10.1002/jcp.10287. PMID 12767050
- [Background] Zhou L, Cai M, Ren Y, Wu H, Liu M, Chen H, Shang J. The different roles of 5-HT1A/2A receptors in fluoxetine ameliorated pigmentation of C57BL/6 mouse skin in response to stress. J Dermatol Sci. 2018 Dec;92(3):222-229. doi: 10.1016/j.jdermsci.2018.10.002. Epub 2018 Oct 25. PMID 30527375
- [Background] Liu L, Fu M, Pei S, Zhou L, Shang J. R-Fluoxetine Increases Melanin Synthesis Through a 5-HT1A/2A Receptor and p38 MAPK Signaling Pathways. Int J Mol Sci. 2018 Dec 25;20(1):80. doi: 10.3390/ijms20010080. PMID 30585252
- [Background] Enkhtaivan E, Lee CH. Role of Amine Neurotransmitters and Their Receptors in Skin Pigmentation: Therapeutic Implication. Int J Mol Sci. 2021 Jul 28;22(15):8071. doi: 10.3390/ijms22158071. PMID 34360837
- [Background] Schallreuter KU, Salem MA, Gibbons NC, Martinez A, Slominski R, Ludemann J, Rokos H. Blunted epidermal L-tryptophan metabolism in vitiligo affects immune response and ROS scavenging by Fenton chemistry, part 1: Epidermal H2O2/ONOO(-)-mediated stress abrogates tryptophan hydroxylase and dopa decarboxylase activities, leading to low serotonin and melatonin levels. FASEB J. 2012 Jun;26(6):2457-70. doi: 10.1096/fj.11-197137. Epub 2012 Mar 13. PMID 22415302
- [Background] Maurer-Spurej E, Dyker K, Gahl WA, Devine DV. A novel immunocytochemical assay for the detection of serotonin in platelets. Br J Haematol. 2002 Mar;116(3):604-11. doi: 10.1046/j.0007-1048.2001.03302.x. PMID 11849219
- [Background] Thompson JH. Iron absorption and serotonin (5-hydroxytryptamine) antagonism. Arch Int Pharmacodyn Ther. 1965 Aug;156(2):249-54. No abstract available. PMID 5868935
- [Background] Amireault P, Hatia S, Bayard E, Bernex F, Collet C, Callebert J, Launay JM, Hermine O, Schneider E, Mallet J, Dy M, Cote F. Ineffective erythropoiesis with reduced red blood cell survival in serotonin-deficient mice. Proc Natl Acad Sci U S A. 2011 Aug 9;108(32):13141-6. doi: 10.1073/pnas.1103964108. Epub 2011 Jul 25. PMID 21788492